CLINICAL TRIAL: NCT01143064
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study to Investigate the Efficacy and Safety of Progesterone in Patients With Severe Traumatic Brain Injury
Brief Title: Efficacy and Safety Study of Intravenous Progesterone in Patients With Severe Traumatic Brain Injury
Acronym: SyNAPSe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BHR Pharma, LLC (Industry)
Collaborators: PRA Health Sciences (Industry); Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHR-100-301; 2010-018283-16 (EudraCT Number)
Record Dates: First submitted 2010-06-10; First posted 2010-06-14 (Estimated); Results first posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Brain Injuries
Keywords: Brain Injury; Trauma
MeSH Terms: conditions — Brain Injuries; Wounds and Injuries | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progesterone (Active Comparator)
  Interventions: Drug: Progesterone
- Lipid emulsion without progestrone (Placebo Comparator)
  Interventions: Drug: Lipid emulsion without progesterone

INTERVENTIONS:
Drug: Progesterone — Intravenous administration of 0.71mg/kg/hr for 1hr followed by 0.5mg/kg/hr administered intravenously for an additional 119 hrs.
  Other Names: BHR-100
  Arms: Progesterone
Drug: Lipid emulsion without progesterone — Intravenous administration equal to 0.71mg/kg/hr for 1hr followed by 0.5mg/kg/hr administered intravenously for an additional 119 hrs.
  Arms: Lipid emulsion without progestrone

SUMMARY:
The SyNAPSe trial will study if giving intravenous (i.v.) progesterone within 8 hours of the injury for a total of 120 hours to severe traumatic brain injury patients improves their recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between the age of 16 and 70 years, inclusive
2. Weight from 45 to 135 kg, inclusive
3. Sustained a closed head trauma no more than 8 hours before start of study drug infusion
4. TBI diagnosed by history and clinical examination
5. Post-resuscitation Glasgow Coma Scale (GCS) score between 3 to 8, inclusive
6. At least one reactive pupil (pinpoint pupils due to opioid pain treatment are considered reactive)
7. Evidence of TBI confirmed by abnormalities consistent with trauma on CT scan upon admission (diffuse injury II-IV, evacuated and non-evacuated mass lesion, Marshall's CT Classification)
8. Indication for ICP monitoring

Exclusion Criteria:

1. Life expectancy of less than 24 hours as determined by the Investigator
2. Prolonged and/or uncorrectable hypoxia (Pa02< 60 mmHg) or hypotension (systolic blood pressure < 90 mmHg) at the time of randomization
3. Any spinal cord injury
4. Pregnancy
5. Penetrating head injury
6. Bilaterally fixed dilated pupils at the time of randomization
7. Coma suspected to be primarily due to other causes (e.g. alcohol)
8. Pure epidural hematoma
9. Preexisting clinically significant disease or chronic condition that can be ascertained at the time of admission and could affect functional outcome
10. Severe cardiac or hemodynamic instability prior to randomization
11. Known treatment with another investigational drug therapy or procedure within 30 days of injury
12. A history of allergic reaction to progesterone and related drugs or any of the components of the infusion
13. Any disease, in the opinion of the Investigator, that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study.
14. Patients who, in the opinion of the Investigator, would not be able or willing to comply with the protocol through the final visit (6 months post-injury)

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1195 (Actual)
Dates: Start 2010-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neta R. Nelson, MPH, Study Director — BHR Pharma, LLC
Locations (156):
- United States (53):
  - University of South Alabama Medical Center, Mobile, Alabama
  - LAC+USC Medical Center, Los Angeles, California
  - University of California San Diego Medical Center, San Diego, California
  - Denver Health Medical Center, Denver, Colorado
  - Christiana Care Health System Hospital, Newark, Delaware
  - Delray Medical Center, Delray Beach, Florida
  - Tallahassee Memorial Healthcare, Tallahassee, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - John H. Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint John's Hospital, Springfield, Illinois
  - Wishard Health Services, Indianapolis, Indiana
  - Methodist Hospital, Indianapolis, Indiana
  - Mercy Medical Center, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville Hospital, Louisville, Kentucky
  - LSU Health - Shreveport, Shreveport, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Medical Center, Portland, Maine
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - St. Mary's of Michigan, Saginaw, Michigan
  - University of Missouri Health Care, Columbia, Missouri
  - Truman Medical Center Hospital Hill, Kansas City, Missouri
  - Lester E. Cox Memorial Hospital, Springfield, Missouri
  - The Nebraska Medical Center, Omaha, Nebraska
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Albany Medical Center Hospital, Albany, New York
  - Westchester Medical Center, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University-Baptist Medical Center, Winston-Salem, North Carolina
  - Summa Health System, Akron, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - St. Elizabeth Health Center, Youngstown, Ohio
  - OU Medical Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital & Health Center, Portland, Oregon
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of South Carolina School of Medicine, Columbia, South Carolina
  - Johnson City Medical Center, Johnson City, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Marshall University Joan C. Edwards School of Medicine, Huntington, West Virginia
  - West Virginia University Hospital, Morgantown, West Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Argentina (7):
  - Hospital Francisco Lopez Lima, General Roca, Río Negro Province
  - Hospital de Emergencias Clemente Alvarez (HECA), Rosario, Santa Fe Province
  - Hospital Nacional "Profesor Alejandro Posadas", Buenos Aires
  - Hospital Regional De Comodoro Rivadavia (HRCR), Comodoro Rivadavia
  - Hospital Central de Mendoza, Mendoza
  - Hospital San Martin, Paraná
  - Hospital Dr. José Maria Cullen, Santa Fé
- Austria (4):
  - Medizinische Universität Graz, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Unfallkrankenhaus Salzburg, Salzburg
  - Landesklinikum Wiener Neustadt, Vienna
- Belgium (5):
  - ULB Erasme, Brussels
  - Ziekenhuis Oost-Limburg, Location Sint Jan, Genk
  - Universitair Ziekenhuis Gent, Ghent
  - University Hospital of the Free University Brussels (UZ Brussel), Jette
  - University Hospital Gasthuisberg, Leuven
- China (8):
  - Chengdu Military General Hospital, Chengdu
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - The 2nd Affiliated Hospital of Zhejiang University, Hangzhou
  - The Second Hospital of Shandong University, Jinan
  - Huashan Hospital of Fudan University, Shanghai
  - Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - General Hospital of Tianjin Medical University, Tianjin
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou
- Czechia (4):
  - Fakultní nemocnice Brno Neurochirurgická klinika, Brno
  - Fakultní nemocnice u sv. Anny v Brnĕ, Neurochirurgická klinika, Brno
  - Fakultní Nemocnice Plzeň, Neurochirurgicé Oddĕlení, Pilsen
  - Fakultní nemocnice Kralovske Vinohrady, Prague
- Tampere University Hospital, Tampere, Finland
- France (8):
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Hôpital Pierre Wertheimer, Bron
  - Centre Hospitalier Universitaire de Grenoble- Hópital Michallon, La Tronche
  - CHRU de Lille- Hópital Roger Salengro, Lille
  - Centre Hospitalier Universitaire de Limoges, Limoges
  - Centre Hospitalier Universitaire Hôpital Nord, Marseille
  - Hópital Central - CHU de Nancy, Nancy
  - Groupe Hospitalier La Salpêtrière, Paris
- Germany (11):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Krankenhaus Merheim, Cologne
  - Klinikum der J.W. Goethe-Universität, Frankfurt
  - Universitätsmedizin Göttingen, Göttingen
  - Berufsgenossenschaftliche Kliniken, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Gießen und Marburg gGmbH, Marburg
  - Klinikum Nürnberg, Nuremberg
  - Niels-Stensen-Kliniken, Osnabrück
  - Universitätsklinikum Ulm, Ulm
- Hungary (3):
  - Honvédelmi Minisztérium Állami Egészségügyi Központ, Budapest
  - Pécsi Tudományegyetem Általános Orvostudományi Kar, Pécs
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
- Israel (5):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Organization, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (6):
  - Fondazione Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena, Milan
  - Fondazione San Raffaele del Monte Tabor, Milan
  - Azienda Ospedaliera San Gerardo, Monza
  - Azienda Ospedaliero Universitaria Maggiore della Caritá, Novara
  - Azienda Ospedaliera San Camillo Forlanini, Rome
  - Azienda Ospedaliero Universitaria Integrata di Verona, Verona
- Malaysia (5):
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Sarawak General Hospital, Kuching
- Netherlands (2):
  - VU Medisch Centrum, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
- Spitalul Clinic Judetean de Urgenta Timisoara, Timișoara, Romania
- Russia (6):
  - State Budget Educational Institution of Higher Professional Education "Kemerovskaya State Medical Academy of Federal Agency of Healthcare and Social Development", Kemerovo
  - State Professional Institution of High Professional Education "Krasnoyarsk State Medical University named after Prof. V.F. Voyno-Yasenetsky of Ministry of Health and Social Development", Krasnoyarsk
  - State Institution "Burdenko Neurosurgical Institute of RAMS", Moscow
  - State Healthcare Facility "Murmansk Regional Clinical Hospital n.a. Bayandin", Murmansk
  - Saint Petersburg Healthcare Institution "City Mariinsky Hospital", Saint Petersburg
  - State Institution of Health Care "Sverdlovsk Regional Clinical Hospital #1", Yekaterinburg
- Singapore (3):
  - National Neuroscience Institute, Singapore
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
- Spain (12):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Parc Taulí, Sabadell, Barcelona
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Universitario Vall Hebrón, Barcelona
  - Hospital Universitario de Girona Dr. Josep Trueta, Girona
  - Hospital Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clínico Universitario De Valencia, Valencia
  - Hospital Universitari i Politecnic La Fé de Valencia, Valencia
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Thailand (3):
  - Chiang Mai University, Chiang Mai
  - Faculty of Medicine, Prince of Songkla University, Hat Yai
  - Khon Kaen Hospital, Khon Kaen
- United Kingdom (7):
  - Royal Preston Hospital, Fulwood, Preston
  - Queen Elizabeth Hospital, Birmingham
  - University Hospital Coventry, Coventry
  - Leeds Teaching Hospitals NHS, Leeds General Infirmary, Leeds
  - The Royal London Hospital, London
  - The James Cook University Hospital, Middlesbrough
  - Southampton University Hospital, Southampton

REFERENCES:
- [Background] Wright DW, Kellermann AL, Hertzberg VS, Clark PL, Frankel M, Goldstein FC, Salomone JP, Dent LL, Harris OA, Ander DS, Lowery DW, Patel MM, Denson DD, Gordon AB, Wald MM, Gupta S, Hoffman SW, Stein DG. ProTECT: a randomized clinical trial of progesterone for acute traumatic brain injury. Ann Emerg Med. 2007 Apr;49(4):391-402, 402.e1-2. doi: 10.1016/j.annemergmed.2006.07.932. Epub 2006 Sep 29. PMID 17011666
- [Background] Xiao G, Wei J, Yan W, Wang W, Lu Z. Improved outcomes from the administration of progesterone for patients with acute severe traumatic brain injury: a randomized controlled trial. Crit Care. 2008;12(2):R61. doi: 10.1186/cc6887. Epub 2008 Apr 30. PMID 18447940
- [Derived] Skolnick BE, Maas AI, Narayan RK, van der Hoop RG, MacAllister T, Ward JD, Nelson NR, Stocchetti N; SYNAPSE Trial Investigators. A clinical trial of progesterone for severe traumatic brain injury. N Engl J Med. 2014 Dec 25;371(26):2467-76. doi: 10.1056/NEJMoa1411090. Epub 2014 Dec 10. PMID 25493978
- See also: Trial website — http://www.synapse-trial.com

RESULTS

PARTICIPANT FLOW:
Groups:
- BHR-100: Progesterone: Intravenous administration of 0.71mg/kg/hr for 1hr followed by 0.5mg/kg/hr administered intravenously for an additional 119 hrs.
- Placebo: Lipid emulsion without progesterone: Intravenous administration equal to 0.71mg/kg/hr for 1hr followed by 0.5mg/kg/hr administered intravenously for an additional 119 hrs.
Period: Overall Study
Arm/Group | BHR-100 | Placebo
Started | 597 | 598
Completed | 464 | 483
Not Completed | 133 | 115
Not completed — Death | 109 | 91
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 7 | 5
Not completed — Lost to Follow-up | 17 | 14
Not completed — Physician Decision | 0 | 4

BASELINE CHARACTERISTICS:
Population: This number is the modified Intention-to-Treat (mITT) Population which includes all subjects who were randomized and in whom treatment with study drug was initiated.
Groups:
- Total: Total of all reporting groups
Arm/Group | BHR-100 | Placebo | Total
Number analyzed (Participants) | 591 | 588 | 1179
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (15.60) | 37.6 (15.36) | 37.4 (15.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 125 | 252
  Male | 464 | 463 | 927
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 61 | 60 | 121
  Not Hispanic or Latino | 479 | 487 | 966
  Unknown or Not Reported | 51 | 41 | 92
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 441 | 458 | 899
  Black/African American/African Heritage | 23 | 16 | 39
  Native Hawaiian/other Pacific Islander | 0 | 0 | 0
  Asian | 63 | 63 | 126
  American Indian or Alaska Native | 2 | 0 | 2
  Not Allowed to Obtain | 51 | 41 | 92
  Other | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  Argentina | 31 | 33 | 64
  Romania | 5 | 1 | 6
  Singapore | 6 | 9 | 15
  Hungary | 3 | 5 | 8
  United States | 219 | 220 | 439
  Czechia | 24 | 34 | 58
  United Kingdom | 24 | 30 | 54
  Malaysia | 11 | 8 | 19
  Thailand | 22 | 24 | 46
  Russia | 6 | 7 | 13
  Spain | 42 | 51 | 93
  Austria | 18 | 14 | 32
  Netherlands | 2 | 5 | 7
  Belgium | 16 | 13 | 29
  China | 20 | 15 | 35
  Finland | 5 | 1 | 6
  Taiwan | 3 | 2 | 5
  Italy | 22 | 24 | 46
  Israel | 37 | 25 | 62
  France | 51 | 41 | 92
  Germany | 24 | 26 | 50
Glasgow Coma Score Motor Score [Count of Participants; unit: Participants] — The Glasgow Coma Scale divides into three parameters: best eye response (E), best verbal response (V) and best motor response (M). The levels of response in the components of the Glasgow Coma Scale are 'scored' from 1, for no response, up to normal values of 4 (Eye-opening response) 5 ( Verbal response) and 6 (Motor response).
  Participants
    1-2 | 129 | 167 | 296
    3 | 84 | 74 | 158
    4 | 167 | 160 | 327
    5-6 | 209 | 185 | 394
    Missing | 2 | 2 | 4
Pupillary Response [Count of Participants; unit: Participants]
  Bilateral | 480 | 475 | 955
  Unilateral | 109 | 107 | 216
  No Reactive Pupils | 0 | 1 | 1
  Not Testable | 2 | 4 | 6
  Missing | 0 | 1 | 1
Hypoxia [Count of Participants; unit: Participants]
  Yes | 15 | 13 | 28
  No | 523 | 521 | 1044
  Suspected | 37 | 32 | 69
  Unknown | 16 | 22 | 38
Hypotension [Count of Participants; unit: Participants]
  Yes | 85 | 66 | 151
  No | 484 | 498 | 982
  Suspected | 8 | 12 | 20
  Unknown | 14 | 12 | 26
Marshall CT Classification [Count of Participants; unit: Participants] — Marshall CT classification of TBI describes 6 categories of severity of TBI based on a non-contrast head CT with binary assessments for presence or absence of:
  1. intracranial abnormalities
  2. CT evidence of increased ICP as demonstrated by a) midline shift (MLS) >5mm and/or
     b) compression of basal cisterns
  3. presence or absence of mass lesions (contusions/hemorrhages)
  4. planned evacuation of mass lesions
  Participants
    I | 6 | 4 | 10
    II | 235 | 233 | 468
    III | 178 | 164 | 342
    IV | 35 | 35 | 70
    Evacuated/Non-Evacuated Mass Lesion | 134 | 151 | 285
    Missing | 3 | 1 | 4
Traumatic Subarachnoid Hemorrhage [Count of Participants; unit: Participants]
  Yes | 449 | 456 | 905
  No | 138 | 131 | 269
  Missing | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Glasgow Outcome Scale (GOS)
Description: The GOS assesses mortality and disability in traumatic brain injury (TBI) patients according to the designation: Good Recovery, Moderate Disability, Severe Disability, Vegetative State or Dead.
Time Frame: 6 months
Population: Only participants with data for this outcome are included. Missing values are first imputed by carrying forward the Month 3 GOS assessment. If a subject has neither the 3 nor the 6 month GOS, the missing value is imputed using the proportional odds model.
Measure: Count of Participants; unit: Participants
Arm/Group | BHR-100 | Placebo
Number analyzed (Participants) | 591 | 588
Participants
  Good Recovery | 189 | 183
  Moderate Disability | 109 | 114
  Severe Disability | 162 | 160
  Vegetative State/Dead | 131 | 131

2. Secondary Outcome: Mortality at Month 1
Description: The mortality rate at one month will be compared between the two treatment groups.
Time Frame: 1 month post injury
Population: P-value population size is based on the number of subjects with status = alive or dead, month 6 within the mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | BHR-100 | Placebo
Number analyzed (Participants) | 591 | 588
Participants
  Lost to Follow-up | 0 | 0
  Consent Withdrawn | 0 | 0
  Alive | 500 | 507
  Dead | 87 | 74
  Other | 1 | 0
  Missing | 3 | 7

3. Secondary Outcome: Mortality at Month 6
Description: The mortality rate at six months will be compared between the two treatment groups.
Time Frame: 6 months post injury
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | BHR-100 | Placebo
Number analyzed (Participants) | 591 | 588
Participants
  Lost to Follow-up | 0 | 2
  Consent Withdrawn | 0 | 0
  Alive | 463 | 472
  Dead | 109 | 95
  Other | 0 | 0
  Missing | 19 | 19

4. Secondary Outcome: Glasgow Outcome Scale at 3 Months
Description: The GOS assesses the mortality and disability in traumatic brain injury patients according to the designation: Good Recovery, Moderate Disability, Severe Disability, Vegetative State, or Dead.
Time Frame: Month 3
Measure: Count of Participants; unit: Participants
Arm/Group | BHR-100 | Placebo
Number analyzed (Participants) | 591 | 588
Participants
  Good Recovery | 103 | 101
  Moderate Disability | 103 | 114
  Severe Disability | 224 | 216
  Vegetative State | 33 | 49
  Dead | 102 | 88
  Missing | 26 | 20

5. Secondary Outcome: Glasgow Outcome Scale - Extended (GOS-E)
Description: The GOS-E assessment of mortality and disability in TBI patients extends the original five GOS categories of functional outcome to eight categories:
  * Dead
  * Vegetative State
  * Lower Severe Disability
  * Upper Severe Disability
  * Lower Moderate Disability
  * Upper Moderate Disability
  * Lower Good Recovery
  * Upper Good Recovery
Time Frame: 3 months and 6 months post injury
Population: Number analyzed (591 for BHR-100 and 588 for placebo) is as listed in the clinical study report. The number analyzed was not modified per time frame and outcome, rather 591 and 588 are included.
Measure: Count of Participants; unit: Participants
Arm/Group | BHR-100 | Placebo
Number analyzed (Participants) | 565 | 568
Participants
  Dead - 3 months | 102 | 88
  Vegetative State - 3 months | 33 | 49
  Lower Severe Disability - 3 months | 173 | 165
  Upper Severe Disability - 3 months | 51 | 51
  Lower Moderate Disability - 3 months | 35 | 34
  Upper Moderate Disability - 3 months | 68 | 80
  Lower Good Recovery - 3 months | 53 | 46
  Upper Good Recovery - 3 months | 50 | 55
  Dead - 6 months: number analyzed (Participants) | 565 | 564
  Dead - 6 months | 109 | 95
  Vegetative State - 6 months: number analyzed (Participants) | 565 | 564
  Vegetative State - 6 months | 20 | 33
  Lower Severe Disability - 6 months: number analyzed (Participants) | 565 | 564
  Lower Severe Disability - 6 months | 115 | 109
  Upper Severe Disability - 6 months: number analyzed (Participants) | 565 | 564
  Upper Severe Disability - 6 months | 37 | 44
  Lower Moderate Disability - 6 months: number analyzed (Participants) | 565 | 564
  Lower Moderate Disability - 6 months | 36 | 38
  Upper Moderate Disability - 6 months: number analyzed (Participants) | 565 | 564
  Upper Moderate Disability - 6 months | 70 | 72
  Lower Good Recovery - 6 months: number analyzed (Participants) | 565 | 564
  Lower Good Recovery - 6 months | 71 | 64
  Upper Good Recovery - 6 months: number analyzed (Participants) | 565 | 564
  Upper Good Recovery - 6 months | 108 | 109

6. Secondary Outcome: Short Form (36) Health Survey (SF-36)
Description: The Short Form (36) Health Survey (SF-36) is a validated survey of patient health consisting of eight scaled scores which are the weighted sums of the questions in their section. The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, role physical, role emotional, role mental and mental health. The maximum score is 30. A score of 23 or lower is indicative of cognitive impairment. The 8 scales can also be further summarized to provide a summary score for physical health and a summary score for mental health. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: 3 months and 6 months post injury
Population: Only participants with data for these parameters have been included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BHR-100 | Placebo
Number analyzed (Participants) | 354 | 369
score on a scale
  Physical Composite Summary - Month 3: number analyzed (Participants) | 332 | 328
  Physical Composite Summary - Month 3 | 39.8 (12.16) | 40.6 (11.37)
  Physical Composite Summary - Month 6 | 44.6 (11.50) | 45.1 (11.30)
  Mental Composite Summary - Month 3: number analyzed (Participants) | 322 | 328
  Mental Composite Summary - Month 3 | 48.7 (12.71) | 48.5 (12.72)
  Mental Composite Summary - Month 6 | 47.9 (11.24) | 46.8 (12.36)

7. Secondary Outcome: Potentially Clinically Important On-Treatment Cerebral Perfusion Pressure (CPP) and Summary of Maximum Therapy Therapeutic Intensity Level (TIL)
Description: Cerebral Perfusion Pressure (CPP) levels are presented according to clinically significant cut-off values. CPP was calculated from intracranial pressures and mean arterial pressures measured from Day through Day 6 after initiation of study medication, if an ICP monitor was in place. Specific therapies received during Days 1-6 are summarized according to the Therapeutic Intensity Level (TIL) by treatment group, as maximum level of therapy administered to the subject.
Time Frame: Admission through post-infusion Day 6
Population: Only participants with data for these parameters have been included.
Measure: Count of Participants; unit: Participants
Arm/Group | BHR-100 | Placebo
Number analyzed (Participants) | 591 | 588
Participants
  Any CPP value < 50 mmHg: number analyzed (Participants) | 531 | 535
  Any CPP value < 50 mmHg | 130 | 155
  Any CPP value >=50-<60 mmHg: number analyzed (Participants) | 531 | 535
  Any CPP value >=50-<60 mmHg | 297 | 299
  Any CPP value >=60-<70 mmHg: number analyzed (Participants) | 531 | 535
  Any CPP value >=60-<70 mmHg | 448 | 460
  Any CPP value >=70 mmHg: number analyzed (Participants) | 531 | 535
  Any CPP value >=70 mmHg | 518 | 523
  Surgical Decompression (TIL) | 192 | 174
  Barbiturate Induced Coma (TIL) | 82 | 73
  Hypothermia (TIL) | 61 | 69
  Hyperventilation (TIL) | 78 | 68
  Pressor Administered (TIL) | 315 | 343
  Hypertonic Saline (TIL) | 225 | 233
  Mannitol (TIL) | 288 | 285
  Ventricular Drainage (TIL) | 198 | 208
  Paralysis Induction (TIL) | 220 | 231
  Sedation (TIL) | 565 | 565

ADVERSE EVENTS:
Arm/Group | BHR-100 | Placebo
All-Cause Mortality (participants affected / at risk) | 109/596 | 95/583
Serious Adverse Events (participants affected / at risk) | 224/596 | 214/583
Other Adverse Events (participants affected / at risk) | 265/596 | 286/583
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BHR-100 (N=596) | Placebo (N=583)
Intracranial pressure increased (Nervous system disorders) | 30 | 27
Brain oedema (Nervous system disorders) | 19 | 17
Hydrocephalus (Nervous system disorders) | 12 | 14
Convulsion (Nervous system disorders) | 9 | 3
Cerebral infarction (Nervous system disorders) | 8 | 5
Pneumonia (Infections and infestations) | 38 | 40
Sepsis (Infections and infestations) | 15 | 14
Septic shock (Infections and infestations) | 11 | 7
Meningitis (Infections and infestations) | 7 | 5
Brain herniation (Injury, poisoning and procedural complications) | 15 | 13
Subdural haematoma (Injury, poisoning and procedural complications) | 10 | 5
Brain contusion (Injury, poisoning and procedural complications) | 5 | 6
Traumatic brain injury (Injury, poisoning and procedural complications) | 4 | 10
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 11
Cardiac arrest (Cardiac disorders) | 7 | 3
Cardio-respiratory arrest (Cardiac disorders) | 6 | 5
Multi-organ failure (Cardiac disorders) | 6 | 7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BHR-100 (N=596) | Placebo (N=583)
Pyrexia (General disorders) | 209 | 229
Hypokalaemia (Metabolism and nutrition disorders) | 94 | 126
Hyperglycaemia (Metabolism and nutrition disorders) | 86 | 85
Hyponatraemia (Metabolism and nutrition disorders) | 59 | 64
Hypophosphataemia (Metabolism and nutrition disorders) | 32 | 49
Hypernatraemia (Metabolism and nutrition disorders) | 39 | 33
Hypomagnesaemia (Metabolism and nutrition disorders) | 32 | 49
Hypocalcaemia (Metabolism and nutrition disorders) | 22 | 29
Hypertension (Vascular disorders) | 129 | 127
Hypotension (Vascular disorders) | 71 | 80
Anaemia (Blood and lymphatic system disorders) | 156 | 159
Thrombocytopenia (Blood and lymphatic system disorders) | 21 | 32
Constipation (Gastrointestinal disorders) | 97 | 102
Gamma-glutamyltransferase increased (Investigations) | 51 | 35
Alanine aminotransferase increased (Investigations) | 30 | 18
Tachycardia (Cardiac disorders) | 69 | 63
Agitation (Psychiatric disorders) | 79 | 78
Diabetes insipidus (Endocrine disorders) | 33 | 43

LIMITATIONS AND CAVEATS:
Treatment Emergent Adverse Events with Incidence of >5% by System Organ Class and Preferred Term (Safety Population) data was reported in the Other (Not Including Serious) Adverse Events section. Adverse events were reported for the modified Intention-to-Treat (mITT) population which includes all subjects who were randomized and in whom treatment with study drug was initiated (analyzed according to randomized treatment).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2011-11-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT01143064/Prot_000.pdf
  • Statistical Analysis Plan (2014-04-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT01143064/SAP_001.pdf